CLINICAL TRIAL: NCT01439256
Title: Telehealth & Remote Measurement Technologies to Improve Medication Adherence in Hypertension
Acronym: HTNMedTrack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Robert H. Friedman, BUMC Faculty, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-28783
Record Dates: First submitted 2011-08-30; First posted 2011-09-23 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer Controlled Telephone Counseling (Experimental): This arm intervenes with subjects and their treating physicians. The intervention is periodic medical adherence promotion counseling for subjects regarding their prescribed HTN medications through a computer-controlled telephone counseling program that has data on subject's recent BP values and their prescribed HTN medications. The subjects' treating physicians receive at regularly scheduled office visits information about subject's recent BP and medication adherence for each prescribed medication and also get physician information and management recommendations
  Interventions: Behavioral: Computer Controlled Telephone Counseling; Other: Physician information and management recommendations
- Usual Care (No Intervention): In this arm, patients with hypertension that is not adequately controlled receive usual care from their physicians. Usual care is defined as receiving regular care from the physician and no additional care or intervention from the study.

INTERVENTIONS:
Behavioral: Computer Controlled Telephone Counseling — The subjects in the intervention arm receive medication adherence counseling through a computer controlled telephone counseling program
  Arms: Computer Controlled Telephone Counseling
Other: Physician information and management recommendations — Treating physicians for those subjects in the intervention arm receive through the medical record system a summary of blood pressure values and adherence data and recommendations.
  Arms: Computer Controlled Telephone Counseling

SUMMARY:
This study focuses on an important patient behavior, medication-taking, and important physician behaviors: promoting medication regimen adherence in patients and appropriately modifying therapy when existing therapy results in inadequate therapeutic effect. The study will also explore the caregivers' (clinicians) behavior after relevant information about their patients' medication adherence and blood pressure control has been provided to them. The investigators focus on behavior change for patients and physicians and seek to change their behaviors to improve the health care delivery process and outcomes. The study aims at facilitating tertiary prevention of cardiovascular, cerebrovascular, and reno-vascular diseases by promoting better blood pressure control.

DETAILED DESCRIPTION:
The study will use state-of-the-art technologies, including two systems that use a telephone-based platform called TLC (Telephone-Linked Care). The two TLC applications have been developed for patients with hypertension (TLC-HTN) as well as patients who have difficulty adhering to their medication regimen (TLC-MED). The investigators will also use state-of-the-art medication monitoring technology (electronic pill trays) that monitor patients' medication-taking behaviors in the intervention and control arms.

The TLC-HTN system was designed for patients with hypertension (HTN) whose blood pressure (BP) was out of control and who were given a home blood pressure monitor. All study subjects (intervention and control) were asked to take their blood pressure at home on a weekly basis. The system gave them feedback on how the reported blood pressure compared to their previous blood pressure values and goals set by their physician. Using self-reported medication-taking behavior provided to the TLC-MED module, TLC-HTN gave the patient additional feedback that linked their adherence to their blood pressure control. At the end of each weekly TLC-HTN conversation, the system sent a report to the patient's physician that displayed recent and previous blood pressure values, identified trends, compared the blood pressures to the physician's goal for the patient and accepted norms, and displayed anti-hypertensive medication use/adherence levels in a similar manner so that the physician could relate adherence to blood pressure control.

TLC-Medication Adherence (TLC-MED): TLC-MED is an additional module that is added to the TLC chronic disease systems including TLC-HTN, with the purpose of promoting medication regimen adherence. In each TLC conversation, TLC-MED will assess the patient's adherence to the medications prescribed for that disease. In this project, the investigators will evaluate two versions of TLC-MED, one which uses an electronic medication event monitoring system to determine medication taking, and the other which uses patient self-report information for determining the same information. The investigators will compare both the self-report method of obtaining medication-taking behavior/adherence and the electronic pill trays to usual care.

Commercially available electronic pill trays for oral, solid medications (e.g., tablets and capsules) will be used by both arms to assess patient medication adherence along with subject self-report of medication-taking. There are a number of methods for conducting medication event monitoring for solid medications. The investigators will use electronic pill trays, consisting of a pillbox containing 28 cups arranged in a 7x4 matrix. Each cup has a sensor that registers when the cup is opened.

ELIGIBILITY:
Inclusion Criteria for Patients:

* A patient at one of the two primary care practices of General Internal Medicine, or in Family Medicine, Boston Medical Center (BMC), whose Primary Care Physician (PCP) is participating in the study.
* A diagnosis of hypertension on the active problem list.
* BP > 140/90 (over 130/80 if diabetic) for two or more consecutive visits (any clinic in the hospital, not limited to PCP but excluding Emergency Department(ED)) over the prior 12 months.
* Having been prescribed at least one anti-hypertension medication (currently listed on the list of prescribed medications).
* Has at least one appointment scheduled with his/her PCP within the next six months.
* Age 18 and over.
* Is planning to continue his/her primary care at Boston Medical Center for at least the next 7 months.
* Is willing and able to use the electronic medication tray unassisted to take the study-selected medication for the next seven months.

Inclusion Criteria for Physicians:

* Be a primary care physician in General Internal Medicine, BMC, or be a primary care physician in Family Medicine, BMC, or be a resident in General Internal Medicine, BMC.
* Have a patient who is eligible and participates in the study.

Exclusion Criteria for Patients:

* Planning to move from the Boston area during the study period.
* No home telephone or touch tone service.
* Cannot use a telephone unassisted.
* Is not willing to receive calls at his/her phone during the study period.
* Does not understand conversational English over the telephone.
* Currently enrolled in the TLC-MultiDisease study.
* Is planning to use another electronic medication tray or bottle (such as Medication Events Monitoring Systems (MEMS) to take the study-selected medication for the next seven months.

Exclusion Criteria for Physicians:

* Not having a patient or patients in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Up to 1 year
  This study will follow the Joint National Committee's (JNC) recommendations for blood pressure. JNC recommends that blood pressure should be reduced to less than 140/90 mm Hg. In this study the investigators will consider blood pressure as a continuous variable and as a binary categorical variable, following the guidelines of the JNC on blood pressure evaluation.

SECONDARY OUTCOMES:
Medication Adherence | Up to 1 year
  Adherence at or over 80% is considered overall medication adherence.
  It is likely that some patient subjects in the intervention group who increase their medication regimen adherence will experience a reduction in their blood pressure. In rare instances, this reduction might lead to a syncopal episode or other medical complications due to hypotension. The investigators expect that such events will be exceedingly rare, yet, possible. TLC is designed to monitor for occurrence of hypotension, and if it occurs, TLC will generate an alert to the patient-subjects' responsible physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Farzanfar, PhD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman RH, Kazis LE, Jette A, Smith MB, Stollerman J, Torgerson J, Carey K. A telecommunications system for monitoring and counseling patients with hypertension. Impact on medication adherence and blood pressure control. Am J Hypertens. 1996 Apr;9(4 Pt 1):285-92. doi: 10.1016/0895-7061(95)00353-3. PMID 8722429
- [Background] King AC, Friedman R, Marcus B, Castro C, Napolitano M, Ahn D, Baker L. Ongoing physical activity advice by humans versus computers: the Community Health Advice by Telephone (CHAT) trial. Health Psychol. 2007 Nov;26(6):718-27. doi: 10.1037/0278-6133.26.6.718. PMID 18020844
- [Background] Kazis LE, Friedman RH. Improving medication compliance in the elderly. Strategies for the health care provider. J Am Geriatr Soc. 1988 Dec;36(12):1161-2. doi: 10.1111/j.1532-5415.1988.tb04406.x. No abstract available. PMID 3192895
- [Background] Friedman RH, Stollerman JE, Mahoney DM, Rozenblyum L. The virtual visit: using telecommunications technology to take care of patients. J Am Med Inform Assoc. 1997 Nov-Dec;4(6):413-25. doi: 10.1136/jamia.1997.0040413. PMID 9391929